CLINICAL TRIAL: NCT00053716
Title: Phase II, Single Center, Non-Controlled, Open-Label Study of Liposomal Prostaglandin E1 (Liprostin) as Adjunct Therapy With Lower Limb Angioplasty in Patients With Ischemic and Non-Ischemic Peripheral Arterial Occlusive Disease
Brief Title: Prostaglandin E1 (Liprostin) Treatment With Lower Limb Angioplasty for Peripheral Arterial Occlusive Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Endovasc (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EV 2002-05; Limb Arterial Disease Study
Record Dates: First submitted 2003-02-04; First posted 2003-02-06 (Estimated); Last update posted 2007-03-07 (Estimated); Status verified 2004-03

CONDITIONS: Peripheral Vascular Disease
Keywords: Angioplasty & PGE1 Treatment of Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

INTERVENTIONS:
Drug: Liprostin [liposomal Prostaglandin E1]

SUMMARY:
This is the first clinical research trial in which intravenous Prostaglandin E1 (PGE1 is a vasoactive hormone) will be used as supportive treatment along with the angioplasty procedure to treat or open up a blocked artery within one lower limb or the most affected of two limbs in subjects with Peripheral Arterial Occlusive Disease.

DETAILED DESCRIPTION:
PAOD results in a decrease in arterial blood flow to the lower limb and feet with symptoms that can include, pain at rest, a numbing sensation in limb or feet, limited ability to walk before pain occurs. PAOD can occur along with diabetic ulcers.

Proposed treatment will be given at a medical center with an overnight hospital stay. Treatment includes angioplasty to open up one or two occluded arteries in a lower limb plus a drug (Liprostin) a special formulation of liposomal Prostaglandin E1,or PGE1, a natural occuring vasoactive hormone). Drug treatment is given twice to each artery to be treated, just before and after angioplasty. When angioplasty procedure is completed, a 12 hour intravenous infusion of Liprostin is given to complete the treatment procedure.

A total of 12 PAOD subjects will be enrolled in a single center: Memorial Hermann Hospital, Houston, TX.

Study will begin in February, 2003 with the last (12th) subject to be enrolled, likely by August, 20

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years and older
* Diagnosis of Peripheral Arterial Occlusive Disease [PAOD]
* Subject is a candidate for immediate angioplasty of the lower limb
* Subject must complete 2 treadmill tests at Screen in which walking distance is limited by PAOD and not due to angina or fatigue

Exclusion Criteria:

* Lower limb peripheral re-vascularization procedures in past 3 months
* History of myocardial infarction in the past 6 months
* Malignant disease, uncontrolled hypertension or Class III heart failure
* Aortic occlusion, thrombosed popliteal aneurysm, severe hemorrhagic disorder, or a long iliac occlusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2003-02; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States